CLINICAL TRIAL: NCT05734651
Title: Prospective Evaluation of the PROMIS Stem for Primary Total Hip Arthroplasty
Brief Title: PROMIS Evaluation Study
Status: Recruiting | Type: Observational
Sponsor: Bezirkskrankenhaus St. Johann in Tirol (Other)
Collaborators: Tyrolean Arthroplasty Registry (Unknown)
Responsible Party: Principal Investigator, Moritz Wagner, Principal Investigator, Bezirkskrankenhaus St. Johann in Tirol
Other Study IDs: 1297/2022
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hip Arthropathy; Osteoarthritis, Hip; Perthes Disease; Osteonecrosis; Femoral Neck Fractures
MeSH Terms: conditions — Osteoarthritis, Hip; Legg-Calve-Perthes Disease; Osteonecrosis; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Intervention
  Interventions: Device: PROMIS Stem

INTERVENTIONS:
Device: PROMIS Stem — Primary Total Hip Arthroplasty with the PROMIS Stem (Fa. Falcon Medical, Mödling, Austria)

SUMMARY:
A total of 250 total hip arthroplasties (THA) are performed at the Bezirkskrankenhaus St. Johann. In a majority of those, implants from the company Falcon Medical (Austria) are used. Those implants are undergoing constant development and improvement. To guarantee their clinical performance, this clinical study is evaluating safety and efficacy of all implants produced by Falcon Medical.

The purpose of this study is to evaluate the effcacy and safety of implants produced and distributed by Falcon Medical. All patients with primary THA and usage of a Falcon Medical implant are included. The outcome measures include intra-operative complications, early post-operative complications, revision for any cause and patient reported outcome (WOMAC questionnaire). All data is prospectively collected in a standardized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty with the PROMIS stem

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient treated with primary total hip arthroplasty at this department are included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2042-02-09 (Estimated)

PRIMARY OUTCOMES:
Stem Migration | 20 years
  Stem Migration measured with the validated EBRA method. The stem migration is assessed in millimeters. The radiograph before surgery and sequential radiographs after surgery are assessed.

SECONDARY OUTCOMES:
WOMAC Score | 20 years
  Patient reported outcome score that is assessed before the surgery and one year after the surgery, 5 years after the surgery, 10 years and 20 years after the surgey.

CONTACTS AND LOCATIONS:
Locations (1):
- BKH St. Johann in Tirol, Department for Orthopedics and Traumatology, Sankt Johann in Tirol, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wagner M, Neururer S, Dammerer D, Nardelli P, Kaufmann G, Braito M, Brunner A. External validation of the Tyrolean hip arthroplasty registry. J Exp Orthop. 2022 Aug 30;9(1):87. doi: 10.1186/s40634-022-00526-3. PMID 36042064